CLINICAL TRIAL: NCT00923377
Title: Pilot Trial to Identify and Characterize Breast Stem Cells in Women at Average Risk and Increased Risk for Breast Cancer
Brief Title: Breast Stem Cells in Women at Average Risk and Increased Risk for Breast Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070123; 07-C-0123; NCT00898105 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-05-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Breast Cancer Prevention; High Risk; Breast Stem Cells; Mammographic Density; Breast Cancer Risk
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Research suggests that breast cancers may arise from a population of stem cells in the normal mammary gland that produce clones of cancer cells.
* Researchers are now trying to determine what events may initiate the formation of cancer cells.

Objectives:

* To look for and describe breast stem cells from normal breast tissue from women who do not have breast cancer.
* To compare the breast stem cells between women at increased risk for breast cancer and women at average risk for breast cancer.
* To show a relationship between the number and type of breast stem cells with the density (appearance) of the mammogram (breast x-ray).
* To make cell cultures (grow cells under controlled conditions) from the breast stem cells.

Eligibility:

-Women 18 years of age and older who are at average or increased risk for breast cancer.

Design:

Participants complete a health history questionnaire, family history questionnaire and risk assessment questionnaire.

* Participants have a mammogram and breast biopsy (surgical removal of a sample of breast tissue).
* Women who can become pregnant have a urine pregnancy test....

DETAILED DESCRIPTION:
Background:

Emerging models of breast cancer suggest that breast cancers arise from a population of stem cells that are present in the normal mammary gland. The stem cell produces a clone of cancer cells.

Researchers are now attempting to isolate and characterize breast stem cells and determine what events may initiate the tumorigenic process.

Objectives:

To identify and characterize breast stem cells from normal breast tissue from women who are free of breast cancer.

To compare characteristics of breast stem cells between women at increased risk for breast cancer and women at average risk for breast cancer.

To correlate breast stem cell number or characteristics with mammographic density.

To establish cell cultures of breast stem cells from women at increased risk for breast cancer and women at average risk for breast cancer.

Eligibility:

Women who are at average or increased risk for breast cancer and over age 18 will be eligible.

Design:

This is a pilot tissue acquisition trial. Breast biopsies will be obtained from all subjects and breast cancer risk demographics will be collected at one time point. We aim to enroll 20 average risk and 20 increased risk women.

ELIGIBILITY:
* INCLUSION CRITERIA:

Women age 18 and older.

No abnormal findings in the breast by physical examination.

Average Risk: must meet all criteria below.

* Gail model index of less than 1.7% over next 5 years.
* Claus model lifetime risk less than 10%.
* BRCAPro and Couch model less than 10% of being a BRCA mutation carrier OR tested negative for documented deleterious BRCA1/2 mutation in family.

Increased risk for invasive breast cancer by one of the following:

* Gail Model risk of greater than 1.7% over 5 years from study entry.
* Claus model lifetime risk to age 79 greater than or equal to 10%.
* History of high risk pathologic lesion: lobular carcinoma in situ, atypical hyperplasia, DCIS (ductal carcinoma in situ).
* Deleterious mutations in BRCA1/2, PTEN or P53.
* Greater than or equal to 10% chance of carrying BRCA1/2 gene mutation as assessed by BRCAPro and Couch model (22, 23). If a woman has a 20% risk of carrying a BRCA1/2 mutation by either model, she will meet eligibility criteria.
* History of unilateral breast cancer either invasive or in situ, and a normal contralateral breast by physical examination.

Willing to stop NSAIDS for 3 days prior to biopsy and aspirin 7 days prior to biopsy.

If history of cancer (other than squamous or basal cell skin cancers), subject must have no evidence of disease at time of enrollment AND no history of cancer directed treatment in the 3 months preceding enrollment.

Identification of dense area of breast tissue suitable for biopsy identified on mammogram by the radiologist.

EXCLUSION CRITERIA:

Current use of hormonal therapies (e.g. tamoxifen, aromatase inhibitors, hormone replacement therapy, oral contraceptive pills, topical or vaginal hormone medications are allowed.)

Chemotherapy and radiation within 3 months prior to breast biopsy procedure.

Breastfeeding within 3 months.

Pregnancy (determined by urine dipstick).

A suspicious unbiopsied lesion by physical examination or mammography of the breast(s) which is being studied.

Bleeding disorder.

Warfarin, low molecular weight heparin, or heparin use.

History of bilateral breast radiation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-03-23; Study Completion 2010-05-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Smith GH, Chepko G. Mammary epithelial stem cells. Microsc Res Tech. 2001 Jan 15;52(2):190-203. doi: 10.1002/1097-0029(20010115)52:23.0.CO;2-O. PMID 11169867
- [Background] Dontu G, Abdallah WM, Foley JM, Jackson KW, Clarke MF, Kawamura MJ, Wicha MS. In vitro propagation and transcriptional profiling of human mammary stem/progenitor cells. Genes Dev. 2003 May 15;17(10):1253-70. doi: 10.1101/gad.1061803. PMID 12756227
- [Background] Kuperwasser C, Chavarria T, Wu M, Magrane G, Gray JW, Carey L, Richardson A, Weinberg RA. Reconstruction of functionally normal and malignant human breast tissues in mice. Proc Natl Acad Sci U S A. 2004 Apr 6;101(14):4966-71. doi: 10.1073/pnas.0401064101. Epub 2004 Mar 29. PMID 15051869